CLINICAL TRIAL: NCT05457192
Title: Glycosylated Hemoglobin and Its Correlations With Electrophysiological Studies and Gait Performance in Diabetic Polyneuropathy Patients
Brief Title: Correlation of HbA1c With Electrophysiological Studies and Gait Performance in Diabetic Polyneuropathy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shereen Saad Eldin Mohamed Ali (Other)
Responsible Party: Sponsor-Investigator, Shereen Saad Eldin Mohamed Ali, Lecturer of physical therapy for Neurology, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/003777
Record Dates: First submitted 2022-07-05; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Diabetic Polyneuropathy
Keywords: Glycosylated hemoglobin; Nerve conduction studies; Diabetic polyneuropathy; Spatiotemporal gait parameters.; Type II DM
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate diabetic polyneuropathy (DPN): 65 patients of both sexes (males & females) with type II DM with moderate polyneuropathy will be included. Patients will be enrolled and assessed for their eligibility to participate in this study. Their body mass index (BMI) will range from 20:30 kg/m2, age will range from 40-60 years, postprandial blood sugar more than 200 mg/dl, duration of diabetic illness five years ago or more and serum Hb1AC will be between 7% and 14%. All the patients suffering from moderate polyneuropathy according to Toronto Clinical Neuropathy Scoring System (TCSS) (score nine to 11 points), and Neuropathy Impairment Score in the lower limbs (NIS-LL) (The muscle power of the lower limbs will be more than grade 2 and less than grade 4)

SUMMARY:
This study will be conducted to investigate the relationship between glycosylated hemoglobin (HbA1c) and nerve conduction studies (NCS) with gait performance in patients with DPN. 65 patients with type II DM with moderate polyneuropathy will participate in this study. Glycosylated Hemoglobin (HbA1c) test will be done for each patient by using the Colorimeter device. Nerve conduction studies (NCS) will be performed for each patient by using the electromyography device to confirm the diagnosis of DPN. The neurophysiological functions of peripheral nerves including (The Common peroneal, Tibial, Sural, and Ulnar motor & sensory branches) will be measured. Spatiotemporal gait parameters (stride length, cadence& velocity) for all the patients will be assessed by two-dimension video-based motion analysis (2D).

DETAILED DESCRIPTION:
The current study is to investigate the correlation between glycosylated haemoglobin (HbA1c) with nerve conduction studies (NCS) including amplitudes, conduction velocities &latency with spatiotemporal gait parameters including stride length, cadence& velocity in patients with diabetic polyneuropathy (DPN). The patients will be recruited from the Out- patient clinic of Faculty of Physical Therapy, Cairo University. All the patients suffering from moderate polyneuropathy according to Toronto Clinical Neuropathy Scoring System (TCSS), and Neuropathy Impairment Score in the lower limbs (NIS-LL). Glycosylated Hemoglobin (HbA1c) test will be done for each patient by using the Colorimeter device. Blood will be collected in a EDTA (3 cm) tube that's attached to the needle. A nerve conduction study will be performed for each patient. Five nerves will be examined in this study including (The common peroneal, tibial, sural and ulnar motor & sensory branches). The Nerve conduction studies involve analysis of specific parameters including amplitude (mv), latency (msec.) and conduction velocity(m/s). The evaluation procedure will be explained to each patient before starting examination. Gait parameters including (stride length, cadence & velocity) will be assessed using 2D video-based motion analysis. The gait will be captured by a digital video camera; (Canon 10 mega pixel - 4x optical zoom, lens 4x15/6.2-24.8mm1:2.7-5.6). The resultant captured film will then be processed using a special software computer program (Adobe premier ver. 6.0).

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis will be confirmed by Nerve Conduction Studies "NCS".
* All the patients suffering from moderate polyneuropathy according to Toronto Clinical Neuropathy Scoring System (TCSS) and Neuropathy Impairment Score (NIS-LL).
* Body mass index (BMI) will range from 20:30 kg/m2.
* Age will range from 40-60 years.
* Postprandial blood sugar more than 200 mg/dl.
* Duration of diabetic illness five years ago or more and serum Hb1AC will be between 7% and 14%.
* Able to walk independently with or without walking aids.

Exclusion Criteria:

* Patients with type I DM.
* History of myopathy or neuromuscular diseases.
* Pregnant females.
* Alcoholics.
* History of major cardiac diseases, heavy metal.
* Other neurological problems as stroke.
* History of ulcers in the lower limbs, foot deformities or malunion fracture of the lower limbs, and acute nerve root compression or advanced arthritis affecting lower extremity.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: This study will include 65 Egyptian patients with type II DM with moderate polyneuropathy. Both sex (males & females) will be included. The patients will be recruited from the Out- patient clinic of Faculty of Physical Therapy, Cairo University. Their body mass index (BMI) will range from 20:30 kg/m2, age will range from 40-60 years, postprandial blood sugar more than 200 mg/dl, duration of diabetic illness five years ago or more and serum Hb1AC will be between 7% and 14%.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
The neurophysiological parameters | At baseline for all patients
  Five nerves will be examined in this study including (The common peroneal, tibial, sural and ulnar motor & sensory branches). Nerve conduction studies (NCS) will be performed by using the electromyography device.
Glycosylated Hemoglobin (HbA1c) level | At baseline for all patients
  Glycosylated Hemoglobin (HbA1c) test will be done for each patient by using the Colorimeter device. The Blood will be collected in a EDTA (3 cm) tube

SECONDARY OUTCOMES:
Spatiotemporal gait parameters | At baseline for all patients
  Spatiotemporal gait parameters for all the patients will be assessed by two-dimension video-based motion analysis (2D).

CONTACTS AND LOCATIONS:
Overall Officials: Shereen Saad Eldin Mohamed, Lecturer, Principal Investigator — lecturer of Neurology at faculty of physical therapy-Cairo university
Locations (1):
- Faculty of physical therapy-Cairo University, Giza, Egypt